CLINICAL TRIAL: NCT03763071
Title: Sleep Patterns and Disturbances in the Second and Third Trimester of Uncomplicated Pregnancy
Brief Title: Sleep Disturbances in the 2nd and 3rd Trimester
Status: Completed | Type: Observational
Sponsor: Bartin State Hospital (Other Government)
Responsible Party: Principal Investigator, Murat Yassa, M.D., Bartin State Hospital
Other Study IDs: 2018-1
Record Dates: First submitted 2018-11-23; First posted 2018-12-04 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Sleep Initiation and Maintenance Disorders; Sleep; Sleep Apnea; Sleep Disorder; Sleep Disturbance; Sleep Apnea, Obstructive; Pregnancy Related; Pregnancy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Apnea Syndromes; Sleep Wake Disorders; Parasomnias; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Pregnant women in the 2nd or 3th trimester Patient-reported scales to measure sleep disorders
  Interventions: Other: Patient-reported scales to measure sleep disorders

INTERVENTIONS:
Other: Patient-reported scales to measure sleep disorders — Patient-reported scales to measure sleep disorders include below mentioned scales:
  Pittsburgh Sleep Quality Index; measures the quality of sleep Berlin Questionnaire; measures the obstructive sleep apnea Stop-Bang questionnaire; measures the obstructive sleep apnea Insomnia Severity Index; measures the insomnia and related parameters

SUMMARY:
Sleep disorders and disturbances are mostly underestimated in clinical practice. Moreover, this problem is generally neglected by the pregnant themselves. Today, it is important to underline any problem that may have an affect to improve the quality of life during pregnancy.

This study assesses the sleep quality, insomnia patterns and obstructive sleep apnea in the second and third trimesters of pregnancy.

DETAILED DESCRIPTION:
Women with uncomplicated pregnancy in the second or third trimester who apply for the routine check will be included.

Specific questionnaires will be used to measure the sleep disorders in addition to the socio-demographic measures:

Pittsburgh Sleep Quality Index, Insomnia Severity Index, Berlin Questionnaire and Stop-Bang Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 2nd or 3rd trimester of pregnancy

Exclusion Criteria:

* Complicated pregnancy
* Multiple pregnancy
* Known sleep disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteered, low-risk, uncomplicated singleton pregnancy
Sampling Method: Probability Sample
Enrollment: 683 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | Through study completion, an average of 39 weeks
  The order of the PSQI items has been modified from the original order in order to fit the first 9 items (which are the only items that contribute to the total score) on a single page. Item 10, which is the second page of the scale, does not contribute to the PSQI score. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Berlin Questionnaire | Through study completion, an average of 39 weeks
  The questionnaire consists of 3 categories related to the risk of having sleep apnea. Patients can be classified into High Risk or Low Risk based on their responses to the individual items and their overall scores in the symptom categories. High Risk: if there are 2 or more categories where the score is positive. Low Risk: if there is only 1 or no categories where the score is positive.
Stop-Bang questionnaire | Through study completion, an average of 39 weeks
  This questionnaire evaluates the risk of sleep apnea. Low risk of OSA: Yes to 0-2 questions Intermediate risk of OSA: Yes to 3-4 questions High risk of OSA: Yes to 5-8 questions or Yes to 2 or more of 4 STOP questions + male gender or Yes to 2 or more of 4 STOP questions + BMI > 35 kg/m2 or Yes to 2 or more of 4 STOP questions + neck circumference.
Insomnia Severity Index (ISI) | Through study completion, an average of 39 weeks
  ISI measures the insomnia and related parameters. Scoring and Interpretation as follows: Add the scores for all seven items (questions 1 + 2 + 3 + 4 + 5 +6 + 7) will give the total score. Total score categories: 0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)

CONTACTS AND LOCATIONS:
Overall Officials: Murat Yassa, MD, Principal Investigator — Bartin State Hospital
Locations (1):
- Bartin State Hospital, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided